CLINICAL TRIAL: NCT01778959
Title: Methods to Manage Intra-operative Floppy-iris Syndrome and Poor Pupil Dilation in Cataract Surgery: an Exploratory Study
Brief Title: Methods to Manage Intra-operative Floppy-iris Syndrome and Poor Pupil Dilation in Cataract Surgery
Acronym: IFIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prim. Univ.-Prof. Oliver Findl, MD, MBA, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IFIS
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Management of Intraoperative Floppy-iris Syndrome and Small Pupils With Different Mechanical Devices

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- standard OVD (Active Comparator)
  Interventions: Device: standard OVD
- Iris hooks (Active Comparator)
  Interventions: Device: Iris hooks
- Malyugin Ring (Active Comparator)
  Interventions: Device: Malyugin Ring
- OVD (Active Comparator)
  Interventions: Device: OVD

INTERVENTIONS:
Device: Malyugin Ring — insertion of a Malyugin Ring to stabilite the pupil during cataract surgery
  Arms: Malyugin Ring
Device: Iris hooks — insertion of iris retractors to stabilize the pupil during cataract surgery
  Arms: Iris hooks
Device: standard OVD — use of a standard cohesive OVD during cataract surgery
  Arms: standard OVD
Device: OVD — use of a highly cohesive OVD during cataract surgery
  Arms: OVD

SUMMARY:
Cataract surgery is one of the most frequently performed surgeries worldwide and complications are rare. However, there are factors that increase the risk of complications, such as poor pupil dilation and intra-operative floppy iris syndrome (IFIS). Reasons for a small pupil size are pseudoexfoliation syndrome (PXF) syndrome, uveitis or synechia and the use of pilocarpin drops. IFIS is a syndrome usually caused by systemic alpha1-blockers (foremost tamsulosin) used to treat benign prostatic hyperplasia.1,2 As described by Chang and Campbell3 IFIS is characterized by billowing of a flaccid iris stroma, a propensity for iris prolapse towards the phacoemulsification tip as well as towards the incisions and progressive intra-operative pupil constriction.

Stopping tamsulosin pre-operatively did not show to effectively prevent IFIS.4,5 However, it is of high importance to identify patients prior to surgery, who are treated with alpha1-blockers, or patients with a small pupil size and poor pharmacological pupil dilation. Some methods, such as intracameral injection of phenylephrine is only sufficient in a few cases 6, and a disadvantage is the risk of a hypertensive episode.7 Another pharmacological method is the use of atropine drops pre-operatively, but this method did not show to sufficiently reduce IFIS.4

Different methods were shown to reduce intra-operative problems due to IFIS/small pupil size:

The use of highly cohesive ophthalmic viscosurgical devices (OVD), also called viscoadaptives, such as sodium hyaluronate (e.g. AMO Healon5 or Croma Eyefill H.D.) help to viscodilate the pupil and by resting on the iris during the entire phacoemulsification procedure reduce the risk of iris prolapsing towards the incisions. This method is more dependent on a central phacoemulsification technique and low fluidic parameters to allow the OVD to stay on the iris during the entire procedure.8 In case of a small pupil, pupil stretching with 2 instruments can be used additively.

Another option to stabilize the pupil size is the use of mechanical pupil expansion devices, such as

1. Iris retractors - these devices are routinely used to dilate the pupil intra-operatively. Typically, 4 or 5 iris retractors, also called iris hooks, are inserted through 4-5 incisions. Usually, the IFIS pupil is very elastic and the risk of overstretching is small.8
2. Pupil expansion rings, such as the Malyugin ring. This ring is placed on the pupil margin with an injector through the main incision. It eliminates the need of additional incisions and saves time.9

Rationale To compare different methods to manage IFIS and poor pupil dilation in cataract surgery: a pupil expansion ring (Malyugin Ring), iris retractors (iris hooks) and a viscoadaptive OVD.

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract
* Age 21 and older
* written informed consent prior to surgery
* Small pupil group: Patients with a pupil size below 4.0 mm after pharmacological dilation with tropicamide 1% and phenylephrine 2.5% gtt as used routinely for pupil dilation,
* IFIS group: Patients, who currently are or have been treated with Alpha-adrenergic receptor antagonists (Tamsulosin- i.e. Alna ret.®)

Exclusion Criteria:

* Pregnancy (pregnancy test will be taken pre-operatively in women of reproductive age)
* Traumatic cataract
* History of uveitis
* Any ophthalmic pathology that could compromise the measurements

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-07 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Mean difference in flare (pre-operatively to 1 day post-operatively) between the OVD and the device group | pre-operatively to 1 day postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, MBA, Principal Investigator — VIROS- Vienna Institute for Research in Ocular Surgery
Locations (1):
- VIROS- Vienna Institute for Research in Ocular Surgery - Department of Ophthalmology, Hanusch Hospital Vienna, Vienna, Vienna, Austria